CLINICAL TRIAL: NCT06139432
Title: Catatonia: Effectiveness of Transcranial Direct Current Electrostimulation (CATATOES)
Acronym: CATATOES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier St Anne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D21-P022
Record Dates: First submitted 2023-11-03; First posted 2023-11-18 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Catatonia
Keywords: transcranial direct-current stimulation; brain stimulation; BFCRS; Chronic catatonia; tDCS; Neurostimulation
MeSH Terms: conditions — Catatonia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active transcranial Direct Current Stimulation (Experimental): Active transcranial Direct Current Stimulation (tDCS): Stimulation of 2mA for 20 minutes
  Interventions: Device: Active tDCS
- Sham transcranial Direct Current Stimulation (Sham Comparator): Sham transcranial Direct Current Stimulation (tDCS): Effective stimulation of 2.5 mA for 30 seconds, then the stimulation stops. The complete session lasts 20 minutes, with 19 minutes and 30 seconds without stimulation.
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: Active tDCS — * Anode opposite the left dorsolateral prefrontal cortex (between F3 and FP1 according to the 10-20 international placement system).
  * Cathode opposite the left temporoparietal junction (between T3 and P3).
  * The stimulation level is 2mA for 20 minutes.
  * Sessions are held twice daily on working days (with a minimum of 3 hours between sessions).
  Twenty sessions will be carried out, two sessions per consecutive working day.
  Other Names: Active transcranial Direct Current Stimulation
  Arms: Active transcranial Direct Current Stimulation
Device: Sham tDCS — * Anode opposite the left dorsolateral prefrontal cortex (between F3 and FP1 according to the 10-20 international placement system).
  * Cathode opposite the left temporoparietal junction (between T3 and P3).
  * Effective stimulation is delivered for 30 seconds (stimulation level is 2 mA), after which effective stimulation stops. The entire session is 20 minutes, with 19 minutes and 30 seconds without stimulation.
  * Sessions are held twice daily on working days (with a minimum of 3 hours between sessions).
  Twenty sessions will be carried out, two sessions per consecutive working day.
  Other Names: Sham transcranial Direct Current Stimulation
  Arms: Sham transcranial Direct Current Stimulation

SUMMARY:
Nearly 10% of people hospitalized in psychiatry have a catatonic syndrome. The treatment of this syndrome is based on lorazepam and electro-convulsive therapy (ECT) in drug-resistant forms. ECT is the reference therapy, very effective in catatonia, but remain difficult to access due to the technical platform required for their realization, leading to delays in the implementation of the treatment responsible for an increase in the morbidity and mortality of catatonia. In this context, a new therapeutic tool available in the treatment of drug-resistant catatonia would improve the prognosis of catatonia. Transcranial direct current stimulation (tDCS) is an alternative, non-invasive brain stimulation technique that does not require anesthesia, and inexpensive and has been shown to be effective in depression and schizophrenia. A series of clinical cases suggests its potential efficacy in catatonia. Our objective is to evaluate the efficacy of tDCS in catatonia in a clinical trial.

DETAILED DESCRIPTION:
Catatonia is a pathology combining affective, motor, behavioural and neuro-vegetative symptoms. Nearly 10% of people hospitalized in psychiatry have a catatonic syndrome. However, it is a severe disorder with a potentially lethal course.

For the treatment of catatonia, lorazepam is effective in most cases, with the percentage of responding patients varying between 70 and 80 per cent, according to the literature. Catatonic episodes resistant to lorazepam are usually associated with chronic catatonia as part of a neurodevelopmental disorder. Genetic abnormalities are often found in these forms of catatonia.

Electroconvulsive therapy (ECT) should be considered for any catatonic episode that is resistant to lorazepam. It is also indicated when a rapid effect must be obtained in life-threatening situations (e.g. malignant catatonia) or when the underlying pathology requires this treatment. Its efficacy is considered excellent, with response rates ranging from 59% to 100%, including when patients have not responded to lorazepam.

There are several limitations to ECT treatment for catatonia:

* There are many centres, particularly in France, where ECT is inaccessible. Delays in access to ECT are particularly acute in rural areas.
* ECT requires a pre-therapeutic assessment, delaying treatment by several days. However, catatonic syndrome is an emergency requiring immediate treatment. Delaying treatment exposes the patient to the risk of aggravation, i.e. malignant catatonia, with a life-threatening outcome.
* ECT treatment is sometimes contraindicated because of contraindications to anaesthesia.

Among neuromodulation techniques, the promising alternative approaches are transcranial magnetic stimulation (rTMS) and transcranial direct current stimulation (tDCS).

Transcranial direct current stimulation (tDCS) is a non-invasive electrical brain stimulation that does not require anaesthesia. The tDCS is based on applying a low direct electrical current (typically less than 20 volts) via two electrodes placed on the scalp. The electric current is applied to the anode (positive electrode) and then flows to the cathode (negative electrode). The electrodes, surrounded by sponges soaked in a saline solution, are positioned at the level of the scalp according to the international 10-20 placement system or, more rarely, according to the MRI-guided neuronavigation system. The device is easily transportable and does not require a specific technical platform.

The present study, randomized versus placebo, aims to test the efficacy of tDCS stimulation on catatonic-resistant syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Men or women over 18 years old
* Under the care of the GHU PARIS Psychiatry and Neurosciences or EPS Ville Evrard.
* Suffering from an episode of catatonia according to the DSM-5 CRITERIA
* Persistence of catatonia criteria according to DSM-5 after 24 hours of lorazepam treatment or contraindication to lorazepam or poor tolerance to lorazepam
* Patient (or guardian) having given informed and written consent
* Beneficiary of a social security plan

Exclusion Criteria:

* Malignant catatonia
* Pregnant or breastfeeding women
* Patients with contraindications to tCDS, namely patients with a defibrillator or a pacemaker, brain stimulator, presence of intracranial metals, uncovered craniectomy or after trepanning.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Bush-Francis Catatonia Rating Scale (BFCRS) | Day 6
  The BFCRS is a comprehensive tool for diagnosing and assessing the severity of catatonic syndrome.
  The BFCRS was devised by Bush, Fink, Petrides, Dowling and Francis in 1996. This scale consists of the assessment of 23 symptoms, scored from 0 to 3. The total score of the BFCRS is the sum of the responses to the 23 items (minimum 0 - maximum 69). High scores reflect a severe disorder.
  Improvement is defined by a 30% decrease in BFCRS scores after 5 days of treatment (10 tDCS sessions)

SECONDARY OUTCOMES:
Bush-Francis Catatonia Rating Scale (BFCRS) | Day 14
  The BFCRS is a comprehensive tool for diagnosing and assessing the severity of catatonic syndrome.
  The BFCRS was devised by Bush, Fink, Petrides, Dowling and Francis in 1996. This scale consists of the assessment of 23 symptoms, scored from 0 to 3. The total score of the BFCRS is the sum of the responses to the 23 items (minimum 0 - maximum 69). High scores reflect a severe disorder.
  The treatment response is assessed as the absolute reduction of the BCRF score after 20 sessions.
Effectiveness of active tDCS vs sham: patients in remission after 20 sessions | every day from Day 1 to Day 14
  Percentage of patients who no longer fulfil the DSM-5 criteria for catatonic syndrome. This criterion was assessed at each session between V1 and V14.
Lorazepam treatment (mg/die) | At baseline then every day from Day 1 to Day 14
  Lorazepam daily administration in mg/die
Percentage of patients requiring electroconvulsive therapy (ECT) | Every day from Day 1 to Day 14
  Percentage of patients requiring electroconvulsive therapy (ECT) during the evaluation period (active vs shamm tDCS)
Occurrence of catatonic syndrome complications | Every day from Day 1 to Day 14
  Pulmonary embolism confirmed by angioscan, transfer to intensive care, pressure sores, inhalation pneumonia requiring antibiotic therapy, death.
To assess the effectiveness of tDCS by comparing changes over time in psychiatric symptomatology: Montgomery-Asberg depression scale (MADRS score) | At baseline, then at Day 1, Day 6, and from Day 11 to Day 14
  The Montgomery-Asberg depression scale (MADRS ) is a 10 -item scale used to assess the severity of depression. High scores reflect a severe disorder (score range 0-60).
To assess the effectiveness of tDCS by comparing changes over time in psychiatric symptomatology: schizophrenia: . Positive and Negative Syndrome Scale (PANSS score) | At baseline, then at Day 1, Day 6, and from Day 11 to Day 14
  PANSS (Positive and Negative Syndrome Scale): is a 30-item scale widely used in schizophrenia research to assess positive and negative psychotic dimensions. The PANSS is composed of 3 subscales: Positive Scale, Negative Scale, and General Psychopathology Scale. Each subscale is rated with 1 to 7 points ranging from absent to extreme. The range for the Positive and Negative Scales is 7-49, and the range for the General Psychopathology Scale is 16-112. The total PANSS score is simply the sum of the sub scales. In addition to these measures, a Composite Scale is scored by subtracting the negative score from the positive score. This yields a bipolar index that ranges from -42 to +42, which is essentially a difference score reflecting the degree of predominance of one syndrome in relation to the other.
To assess the effectiveness of tDCS by comparing changes over time in psychiatric symptomatology: hypomanic or manic episode: Young Mania Rating Scale (YMRS score) | At baseline, then at Day 1, Day 6, and from Day 11 to Day 14
  The Young Mania Rating Scale (YMRS) is a rating scale used to evaluate manic symptoms : there are eleven items, each item given a severity rating. Four are graded on a 0 to 8 scale (irritability, speech, thought content, and disruptive/aggressive behavior), while the remaining seven items are graded on a 0 to 4 scale.High scores reflect a severe disorder (score range 0-60)
Evolution of physiological parameters: Electrocardiography (ECG) | Baseline then every day from Day 1 to Day 14
  ECG values for waves and intervals: RR interval(seconds);P wave (milliseconds); PR (milliseconds);PR segment (milliseconds); QRS complex (milliseconds) ;ST segment (milliseconds); T wave:(milliseconds) ;QT interval (milliseconds )
Evolution of physiological parameters: blood pressure (systolic pressure and a diastolic pressure mm HG) | Baseline then every day from Day 1 to Day 14
  Blood pressure (systolic pressure and a diastolic pressure mm HG)
Evolution of physiological parameters: brething system | Baseline then every day from Day 1 to Day 14
  Brething system: breaththig freaquency ( breath per minute);
Evolution of physiological parameters: Body temperature °C | Baseline then every day from Day 1 to Day 14
  Body temperature °C
Evolution of physiological parameters: Skin conductance level (SCL) | Baseline then every day from Day 1 to Day 14
  Skin conductance level (SCL value μS)

CONTACTS AND LOCATIONS:
Overall Officials: Marion Plaze, MD,PHD, Study Chair — Groupe Hospitalier Universitaire (GHU) Psychiatrie et Neurosciences; Alexandre Haroche, MD,PHD, Principal Investigator — Groupe Hospitalier Universitaire (GHU) Psychiatrie et Neurosciences
Locations (2):
- France (2):
  - CRC Pôle 93G03 Etablissement Public de Santé EPS Ville Evrard, Neuilly-sur-Marne, Île-de-France Region
  - Groupe Hospitalier Universitaire (GHU) Psychiatrie et Neurosciences, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sienaert P, Dhossche DM, Vancampfort D, De Hert M, Gazdag G. A clinical review of the treatment of catatonia. Front Psychiatry. 2014 Dec 9;5:181. doi: 10.3389/fpsyt.2014.00181. eCollection 2014. PMID 25538636
- [Background] Solmi M, Pigato GG, Roiter B, Guaglianone A, Martini L, Fornaro M, Monaco F, Carvalho AF, Stubbs B, Veronese N, Correll CU. Prevalence of Catatonia and Its Moderators in Clinical Samples: Results from a Meta-analysis and Meta-regression Analysis. Schizophr Bull. 2018 Aug 20;44(5):1133-1150. doi: 10.1093/schbul/sbx157. PMID 29140521
- [Background] Sarkar S, Sakey S, Mathan K, Bharadwaj B, Kattimani S, Rajkumar RP. Assessing catatonia using four different instruments: Inter-rater reliability and prevalence in inpatient clinical population. Asian J Psychiatr. 2016 Oct;23:27-31. doi: 10.1016/j.ajp.2016.07.003. Epub 2016 Jul 11. PMID 27969074
- [Background] Hawkins JM, Archer KJ, Strakowski SM, Keck PE. Somatic treatment of catatonia. Int J Psychiatry Med. 1995;25(4):345-69. doi: 10.2190/X0FF-VU7G-QQP7-L5V7. PMID 8822386
- [Background] Haroche A, Giraud N, Vinckier F, Amad A, Rogers J, Moyal M, Canivet L, Berkovitch L, Gaillard R, Attali D, Plaze M. Efficacy of Transcranial Direct-Current Stimulation in Catatonia: A Review and Case Series. Front Psychiatry. 2022 Apr 27;13:876834. doi: 10.3389/fpsyt.2022.876834. eCollection 2022. PMID 35573356
- [Background] Moyal M, Plaze M, Baruchet A, Attali D, Cravero C, Raffin M, Consoli A, Cohen D, Haroche A, Chaumette B. Efficacity of tDCS in catatonic patients with Phelan McDermid syndrome, a case series. Brain Stimul. 2022 Nov-Dec;15(6):1432-1434. doi: 10.1016/j.brs.2022.10.005. Epub 2022 Oct 26. No abstract available. PMID 36309344